CLINICAL TRIAL: NCT03761966
Title: Cytokines Profile at the Beginning of Pregnancy in Mexican Women
Brief Title: Cytokines Profile at the Beginning of Pregnancy
Status: Completed | Type: Observational
Sponsor: Materno-Perinatal Hospital of the State of Mexico (Other)
Collaborators: Universidad Autonoma del Estado de Mexico (Other); Ciprés Grupo Médico CGM SC (Other)
Responsible Party: Principal Investigator, Hugo Mendieta Zeron, Chief of the Research Department, Materno-Perinatal Hospital of the State of Mexico
Other Study IDs: 217B500402015066
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Correlation of Cytokines and Anthropometry in Pregnancy
Keywords: IL-10; IL-4; IFN-γ; TNF-α; Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women older than 18 years old atended at the "Mónica Pretelini Sáenz" Maternal-Perinatal Hospital (HMPMPS), Health Institute of the State of Mexico (ISEM).
  Interventions: Other: Pregnant women

INTERVENTIONS:
Other: Pregnant women

SUMMARY:
A mechanism by which obesity could influence the increase in obstetric complications as more weight is gained, apart from oxidative stress (3) would be the changes in the expression profile of T helper (Th) cells. Due to the increase rate of obesity among Mexican women, the aim was to determine if there is some association between the weight changes in pregnancy and the cytokines Interleukin (IL)-10, IL-4, Interferon gamma (IFN-γ) and Tumor Necrosis Factor alpha (TNF-α).

DETAILED DESCRIPTION:
Pregnant women older than 18 years old were invited to participate and all were asked to sign the informed consent. Women with congenital heart disease, disabling diseases, infectious diseases and autoimmune diseases were excluded and those whose clinical follow-up was lost were discarded from the final analysis.

Weight and height were measured using a calibrated using an adult scale (Seca, Hamburg, Germany). Blood Pressure (BP; mmHg) was checked by auscultation using a standard sphygmomanometer (Riester Big Ben® Square; Jangingen, Germany). All mothers received written nutritional guidance depending on the characteristics of each patient.

The expression levels of IL-10, IL-4, IFN-γ and TNF-α was performed by the ELISA technique.

Quantitative variables will be represented by measures of central tendency. Once the Kolmogorov test is performed for the normality of the variables, either the Student's T test or the Mann Whitney U test will be used to compare both groups. With the same criteria for normality either Pearson or Spearmen correlation will be used among the cytokines and anthropometric variables, considering a significant difference at p ≤ 0.05. The statistical analysis will be carried out in the Statistical Package for the Social Sciences (SPSS) program, version 19.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women older than 18 years old were invited to participate and all were asked to sign the informed consent.

Exclusion Criteria:

* Women with congenital heart disease, disabling diseases, infectious diseases and autoimmune diseases were excluded and those whose clinical follow-up was lost were discarded from the final analysis.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women.
Study Population: Pregnant women older than 18 years old attender at the "Mónica Pretelini Sáenz" Maternal-Perinatal Hospital, located in Toluca City.
  For a population of 8500 pregnant women annually attended, and a margin of error of 11%, the sample should be of 79 people.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Cytokines levels | 2017-2018
  The expression levels of IL-10, IL-4, IFN-γ and TNF-α will be performed by the ELISA technique on an ELx800 ™ device (BioTek Instruments, Inc.) at the Research Laboratory of Ciprés Grupo Médico S.C. (CGM).

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Mendieta Zerón, PhD, Principal Investigator — Maternal-Perinatal Hospital "Mónica Pretelini Sáenz"
Locations (1):
- Materno-Perinatal Hospital "Mónica Pretelini", Toluca, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
The final data will be available upon request if requiered by the selected journal to publish the final manuscript.

REFERENCES:
- [Background] Lombardelli L, Aguerre-Girr M, Logiodice F, Kullolli O, Casart Y, Polgar B, Berrebi A, Romagnani S, Maggi E, Le Bouteiller P, Piccinni MP. HLA-G5 induces IL-4 secretion critical for successful pregnancy through differential expression of ILT2 receptor on decidual CD4(+) T cells and macrophages. J Immunol. 2013 Oct 1;191(7):3651-62. doi: 10.4049/jimmunol.1300567. Epub 2013 Aug 30. PMID 23997222
- [Background] Cheng SB, Sharma S. Interleukin-10: a pleiotropic regulator in pregnancy. Am J Reprod Immunol. 2015 Jun;73(6):487-500. doi: 10.1111/aji.12329. Epub 2014 Oct 1. PMID 25269386
- [Background] Ziganshina MM, Krechetova LV, Vanko LV, Nikolaeva MA, Khodzhaeva ZS, Sukhikh GT. Time course of the cytokine profiles during the early period of normal pregnancy and in patients with a history of habitual miscarriage. Bull Exp Biol Med. 2013 Jan;154(3):385-7. doi: 10.1007/s10517-013-1956-0. PMID 23484206
- [Background] Wegmann TG, Lin H, Guilbert L, Mosmann TR. Bidirectional cytokine interactions in the maternal-fetal relationship: is successful pregnancy a TH2 phenomenon? Immunol Today. 1993 Jul;14(7):353-6. doi: 10.1016/0167-5699(93)90235-D. PMID 8363725